CLINICAL TRIAL: NCT01754025
Title: INHERIT EGFR - INvestigating HEreditary RIsk From T790M: A Multi-Centered Study to Identify and Characterize Individuals Carrying Germline EGFR Mutations
Brief Title: INHERIT EGFR - Studying Germline EGFR Mutations
Acronym: INHERIT
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Principal Investigator, Jaclyn LoPiccolo, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 12-360
Record Dates: First submitted 2012-12-17; First posted 2012-12-21 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Gene Mutation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cancer patients with T790M: Have a diagnosis of cancer of any type. Have an EGFR T790M mutation identified on either genotyping of their cancer at diagnosis OR on quantitative plasma genotyping with evidence of high level (>40% allelic fraction) EGFR T790M. OR another EGFR mutation previously reported as germline detected on tumor genotyping of their cancer.
- Relatives of Carriers: Have a relative known to carry a germline EGFR mutation (either T790M or other novel germline EGFR mutation)
- Individuals known to be carriers: Have a known germline EGFR mutation (either T790M or other novel germline EGFR mutation)

SUMMARY:
Lung cancer is a common malignancy that is associated with cigarette smoking but can also affect individuals who never smoked. It is not well understood whether there are hereditary risk factors that influence the risk of lung cancer.

It has been recently found that a small number of families have an inherited (passed from parent to child) change in one of their genes that may contribute to an increased tendency to develop lung cancers, even in never smokers. In some lung cancer patients this gene, called "EGFR", contains a DNA change known as an "inherited EGFR mutation". Early data indicate that these inherited EGFR mutations may be associated with an increased risk of lung cancer.

So far, only a small number of families have been found to carry inherited EGFR mutations. For this reason the risk of lung cancer associated with inherited EGFR mutations is not well understood. Understanding the risk may help investigators find ways of detecting lung cancer sooner or reducing the risk of developing lung cancer.

It was recently discovered that lung cancer patients who are found to carry one rare EGFR mutation in their cancer cells, called "T790M", have an increased risk of carrying an inherited EGFR mutation in their normal cells as well. This represents a new strategy for finding individuals and families carrying inherited EGFR mutations.

This research study is designed to find cancer patients whose tumors have this EGFR mutation, T790M, to find out if they also have an inherited EGFR mutation. Subjects will not have to undergo a biopsy to participate in this research study. Investigators will collect a saliva specimen from patients with a T790M in their cancer to find out if they also have an inherited EGFR mutation.

Study participants found or known to carry an inherited EGFR mutation will have the option of offering their close relative the opportunity to also participate in this study. Close relatives can consider testing to see if they also carry the inherited mutation in their normal cells. Once investigators have identified individuals and relatives that carry inherited EGFR mutations in their genes, investigators will then try to understand the risk of lung cancer and other cancers. Individuals with inherited EGFR mutations will also have the opportunity to participate in future studies related to cancer and other diseases.

This study is being funded in part by the Conquer Cancer Foundation of ASCO and the Bonnie J. Addario Lung Cancer Foundation.

DETAILED DESCRIPTION:
If a subject have lung cancer or another cancer carrying a T790M mutation in the EGFR gene, he/she may be eligible to participate in this research study. To determine eligibility, a subject will need to perform the following steps: provide informed consent, fill out the study questionnaire and provide medical records documentation.

The study questionnaire should take about 30 minutes to complete. The questionnaire asks for information on personal and family cancer and health history. The information provided will help investigators to determine which parts of the study a subject is eligible for. A few weeks after submitting the questionnaire, a member of the research study team will contact the subject by telephone to clarify any questions about the response.

For medical records documentation investigators will request permission to obtain and review medical records pertaining to any personal history of cancer. Subjects will need to complete a medical record release form to allow investigators to collect medical records regarding prior cancers and cancer treatment.

After a subject is determined to be eligible, he/she will have a conversation with a genetic counselor regarding the potential risks, benefits and limitations of genetic testing. A genetic counselor is an expert in the field of inherited disorders. They work as members of the health care team and act as a patient advocate providing education and support to the patient, family and the medical team. If a subject agrees to proceed, he/she will be provided a kit (by mail or in person) to provide a saliva sample for genetic testing. This involves spitting into a special container provided by the study. This sample will be sent to a clinically-certified testing laboratory to determine presence of an inherited EGFR mutation.

Once the results have been determined, the subject will receive a letter with the phone number of a genetic counselor to call in order to review results of the genetic testing. Alternatively, a subject can decide not to receive the results of the genetic testing and can note that on the letter received and send it back to the study team instead of calling for the results.

If a mutation is found in the saliva sample, a subject will receive information about how to undergo confirmatory testing of a blood specimen. This can be done at a local laboratory using a kit that will be mailed. When the results are available a genetic counselor will call to discuss them. If the confirmatory blood test confirms an inherited mutation, subjects will receive instructions on how to invite family members to be tested if appropriate.

Investigators will collect material from a prior tumor biopsy (if available), copies of imaging scans, and medical records to study. The copies of imaging scans will allow study of the characteristics of nodules in the lungs. This information will be used to answer additional questions about cancers carrying EGFR T790M mutations.

It will only take a few months to complete the main part of the study. After that, subjects will be followed every 6 months for 2 years. If a subject allows a piece of a tumor specimen or DNA to be stored for future investigational studies, then he/she will remain enrolled in research for as long as the specimen is stored in the specimen bank.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study a subject must meet the eligibility of one of the following cohorts:

Cohort 1 - Cancer patients with T790M in their tumor must both:

* Have a diagnosis of cancer of any type (lung cancer or other)
* Have an EGFR mutation identified. Either EGFR T790M identified on tumor genotyping of their cancer OR on quantitative plasma genotyping with evidence of high level (>40% allelic fraction) EGFR T790M OR
* Another EGFR mutation previously reported as germline detected on tumor genotyping of their cancer

Cohort 2 - Relatives of carriers of germline EGFR mutations are eligible as follows:

* First-degree or second-degree relatives of an individual known to carry a germline EGFR mutation (either T790M or other novel germline EGFR mutation)
* Third-degree relatives of an individual known to carry a germline EGFR mutation (either T790M or other novel germline EGFR mutation) if the relative has a personal history of lung cancer or another malignancy

Cohort 3 - Individuals already known to carry a germline EGFR mutation must:

* Have a known germline EGFR mutation (either T790M or other novel germline EGFR mutation)

Exclusion Criteria:

* Subjects with lung cancer and an acquired T790M mutation first detected after exposure to an EGFR tyrosine kinase inhibitor such as erlotinib or gefitinib
* Subjects who are too ill to complete the study questionnaire or provide the necessary specimen for testing
* Subjects who are unable to give informed consent
* Subjects who are unable to speak or read English or Brazilian Portuguese
* Subjects under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified through participating cancer centers as well as a study website (www.dana-farber.org/T790Mstudy)
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-12-28 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of EGFR mutations | 2 years
  To determine the prevalence of germline EGFR mutations in lung cancer patients with EGFR T790M mutations in their tumor and in relatives of carriers of germline EGFR mutations

SECONDARY OUTCOMES:
Preliminary Assessment of History of Lung Cancers | 2 years
  To make a preliminary assessment of the natural history of lung cancers occurring in patients with germline EGFR mutations
Estimate of Prevalence of Lung Nodules | 2 years
  To generate an initial estimate of the prevalence of CT-detected lung nodules in individuals with germline EGFR mutations
Study EGFR Expression in Skin Biopsies | 2 years
  To study EGFR expression in skin biopsies from patients on study
Explore Relationship Between High Allelic Fraction T790M in plasma genotyping and germline mutations | 2 years
  To explore the relationship between high allelic fraction T790M on plasma genotyping and presence of an underlying germline EGFR T790M mutation
Examine Lung Cancer Risk Associated with Other Germline Mutations | 2 years
  To study individuals and families with rare germline mutations, such as EGFR V843I and EGFR R776H

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn LoPiccolo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Background] Oxnard GR, Miller VA, Robson ME, Azzoli CG, Pao W, Ladanyi M, Arcila ME. Screening for germline EGFR T790M mutations through lung cancer genotyping. J Thorac Oncol. 2012 Jun;7(6):1049-52. doi: 10.1097/JTO.0b013e318250ed9d. PMID 22588155
- [Derived] Oxnard GR, Chen R, Pharr JC, Koeller DR, Bertram AA, Dahlberg SE, Rainville I, Shane-Carson K, Taylor KA, Sable-Hunt A, Sholl LM, Teerlink CC, Thomas A, Cannon-Albright LA, Fay AP, Ashton-Prolla P, Yang H, Salvatore MM, Addario BJ, Janne PA, Carbone DP, Wiesner GL, Garber JE. Germline EGFR Mutations and Familial Lung Cancer. J Clin Oncol. 2023 Dec 1;41(34):5274-5284. doi: 10.1200/JCO.23.01372. Epub 2023 Oct 23. PMID 37579253